CLINICAL TRIAL: NCT02253732
Title: Skeletal Muscle as a Mediator of Exercise Induced Effects on Metabolism & Cognitive Function: Role for Myokines & miRNAs
Acronym: Brain-Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Slovak Academy of Sciences (Other Government)
Collaborators: University Hospital Bratislava (Other)
Responsible Party: Principal Investigator, Jozef Ukropec, PhD, Slovak Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UEE-SAS
Record Dates: First submitted 2014-09-25; First posted 2014-10-01 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Parkinson Disease; Healthy Volunteers
Keywords: MicroRNAs; exercise; skeletal muscle; metabolism
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Parkinson Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- '3 months exercise intervention program' (Experimental): all participants will be subjected to 3 months supervised exercise intervention programme
  Interventions: Behavioral: 3 months exercise intervention program

INTERVENTIONS:
Behavioral: 3 months exercise intervention program — 3 months exercise intervention program which is given 3-times per week, 60 min session duration, 65-75% repetition maximum or heart rate maximum, combined strength & aerobic exercises

SUMMARY:
The purpose of this study is to determine specific changes in muscle secretory profile (myokines, miRNA) in association with neurodegenerative disease progression and metabolic dysfunction. Next the investigators would like to determine the shift in the muscle secretory activity induced by regular exercise intervention, which the investigators think could be translated into the beneficial changes in clinical phenotypes, determined by neuroimaging, cognitive function tests and metabolic phenotyping.

DETAILED DESCRIPTION:
Standard Operating Procedures for patient recruitment, data collection, data management, data analysis routinely used in University Hospital Bratislava and in Institute of Experimental Endocrinology Slovak Academy of Sciences will be employed.

Statistical analysis will be employed to address the primary and secondary objectives, as specified in the study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Diagnosed with Parkinson disease
3. Diagnosed with mild cognitive impairment (MCI) or Alzheimer disease (AD)

Exclusion Criteria:

1. Serious systemic cardiovascular, hepatic, renal disease, cancer.
2. Lack of compliance.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
muscle microRNAs and myokines | up to 24 months
  We will determine muscle bioactive secretory products (myokines & miRNAs) that are regulated by acute bout of exercise in patients with neurodegenerative disease as well as in sedentary age, gender and BMI matched controls in association with their metabolic phenotype.
whole body energy metabolism | up to 24 months
  changes in whole body energy metabolism will be determined with indirect calorimetry. & oral glucose tolerance test
cognitive function | up to 24 months
  exercise related changes in cognitive & motoric functions will be determined with the aid of questionaires, and proton (1H)-magnetic resonance spectroscopy - brain imaging and spectroscopy
motoric function | up to 30 months
  Proton (1H)-magnetic resonance spectroscopy - brain imaging and spectroscopy, motoric - balance testing

SECONDARY OUTCOMES:
Muscle functional tests | up to 30 months
  Dynamometry will be used to determine maximal voluntary contraction force and the rate of force development, and Phosphorus (31P)-magnetic resonance spectroscopy to measure muscle metabolism in vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Valkovic, MD, PhD, Study Chair — University Hospital Bratislava; Stanislav Sutovsky, MD, PhD, Study Chair — University Hospital Bratislava
Locations (2):
- Slovakia (2):
  - Univeristy Hospital in Bratislava, Bratislava
  - Inst. Exp. Endocrinology Slovak Acad Sci, Bratislava

REFERENCES:
- [Derived] Krumpolec P, Vallova S, Slobodova L, Tirpakova V, Vajda M, Schon M, Klepochova R, Janakova Z, Straka I, Sutovsky S, Turcani P, Cvecka J, Valkovic L, Tsai CL, Krssak M, Valkovic P, Sedliak M, Ukropcova B, Ukropec J. Aerobic-Strength Exercise Improves Metabolism and Clinical State in Parkinson's Disease Patients. Front Neurol. 2017 Dec 22;8:698. doi: 10.3389/fneur.2017.00698. eCollection 2017. PMID 29312123